CLINICAL TRIAL: NCT05700916
Title: Evaluation of Milk Polar Lipids on Lipoprotein Metabolism, Inflammation, and Gut Microbiota in Dyslipidemic Adults With Abdominal Obesity
Brief Title: Evaluation of Milk Polar Lipids in Dyslipidemic Adults With Abdominal Obesity
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Blesso, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H22-0161
Record Dates: First submitted 2023-01-10; First posted 2023-01-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Dyslipidemias; Obesity
MeSH Terms: conditions — Dyslipidemias; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MPL-rich dairy powder (Experimental): Daily consumption of 50 g of dairy powder containing 6.5 g MPL for 8 weeks.
  Interventions: Drug: Milk Polar Lipid-Rich Dairy Powder
- Control dairy powder (Placebo Comparator): Daily consumption of 50 g of dairy powder containing <0.1 g MPL for 8 weeks
  Interventions: Dietary Supplement: Dairy Powder

INTERVENTIONS:
Drug: Milk Polar Lipid-Rich Dairy Powder — Effects of the addition of 6.5 g of milk polar lipids to dairy powder.
  Arms: MPL-rich dairy powder
Dietary Supplement: Dairy Powder — Effects of dairy control powder
  Arms: Control dairy powder

SUMMARY:
The major objective of this project is to examine whether daily consumption of milk polar lipids (MPLs) influences cardiometabolic risk factors.

DETAILED DESCRIPTION:
The investigators will conduct a randomized, double-blind, controlled, parallel, intervention study in dyslipidemic adults with abdominal obesity (n = 130). Participants will consume either a control dairy beverage (n = 65) or an MPL-rich dairy beverage (n = 65) for 8 weeks. The investigators plan to evaluate the following 4 specific objectives:

1. Determine the effects of MPLs on serum lipid concentrations and other cardiometabolic risk factors.
2. Evaluate the effects of MPLs on systemic biomarkers of low-grade inflammation.
3. Examine the effects of MPLs on lipoprotein metabolism and lipoprotein particle characteristics.
4. Evaluate the effects of MPLs on gut microbiota, gut permeability markers, and fecal lipids.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C ≥ 130 mg/dL
* Waist circumference ≥ 88 cm for women, ≥ 102 cm for men
* Aged 18 to 70 years

Exclusion Criteria:

* Renal disease
* Liver disease
* Diabetes
* Heart disease
* Stroke
* Cancer
* Eating disorders
* Thyroid disease
* Gut-associated pathologies
* Autoimmune diseases
* Chronic inflammatory diseases
* Scleroderma
* Gallbladder disease
* Blood clotting disorders
* Intravenous drug use
* Fasting plasma/serum triglycerides >500 mg/dL
* Fasting plasma/serum glucose >126 mg/d
* Weight changes >10% over last 4 weeks
* Oral antibiotics use up to 1 month prior to and during study
* Allergy or intolerance to milk products
* Taking lipid-lowering medications (e.g., statins, fibrates)
* Taking anti-inflammatory medications (e.g., corticosteroids)
* Taking medications which primarily affect blood clotting (e.g., warfarin).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Serum LDL Cholesterol at 8 weeks | 8 weeks
  Measurement of serum LDL cholesterol (mg/dL) at the beginning and end of 8-week intervention arm.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States